

# **Study Protocol**

| Title: | Prevalence of cardiovascular disease in Swedish patients with type 2 diabetes and in patients initiating on Empagliflozin (ATC code A10BK03) |
|---|---|
| Study code | F_07_2018 |
| Responsible statistician: | |
| Responsible project epidemiologist: | |
| Date of Study<br>Protocol: | 22-Feb-2018 |
| Version: | 0.2 |
| | Page 1 of 10 |

# Table of Contents

| List of abbreviations | 3 |
|----------------------------------------------|----|
| Introduction | 4 |
| Research question and objectives | 5 |
| Research questions | 5 |
| Objectives | 5 |
| Primary objectives | 5 |
| Secondary objectives | 5 |
| Subject sets analyzed | 5 |
| Source population in the study | 5 |
| Index date | 6 |
| Baseline and look back period | 6 |
| Established CVD | 6 |
| Initiation on Empagliflozin | 7 |
| Other variables | 7 |
| Demographics and clinical baseline variables | 7 |
| Planned analysis | 9 |
| Summary of study populations identification | 9 |
| Main analysis | 9 |
| Data management | 9 |
| Statistical software. | 10 |
| Quality control | 10 |
| References | 10 |

# List of abbreviations

| Term | Definition / description |
|--------|------------------------------------------|
| BMI | Body mass index |
| CDR | Cause-of-Death register |
| CI | Confidence interval |
| eGFR | Estimated glomerular filtration rate |
| HbA1c | Glycated haemoglobin A1c |
| HDL | High Density Lipoprotein |
| ICD-10 | International classification of diseases |
| MI | Myocardial infarction |
| NDR | National diabetes register |
| NPR | National patient register |
| PH | Proportional hazards |
| PS | Propensity score |
| RR | Relative risk |
| SPDR | Swedish prescribed drug register |
| T1DM | Type 1 diabetes mellitus |
| T2DM | Type 2 diabetes mellitus |
| | • • |

#### Introduction

The Swedish National Diabetes Register (NDR) was launched in 1996 for the purpose of promoting evidence-based development of diabetes care. The NDR has been online since April 2002 (www.ndr.nu), allowing individual clinics to quickly monitor their activities on a regular basis. The register offers a unique opportunity to monitor the quality of care in terms of risk factors and the potential complications of diabetes. The results generated by the register have been presented at many international meetings and conferences. To our knowledge, the NDR is the largest diabetes register in the world.

Patients with Type 2 diabetes mellitus (T2DM) are at high risk for developing cardiovascular disease (CVD) complications.

The EMPA-REG OUTCOME (ERO) trial demonstrated a reduction in cardiovascular death, hospitalization from heart failure and all-cause mortality. Empagliflozin also reduces the risk for new onset or worsening of nephropathy, progression to macroalbuminuria and doubling of serum creatinine accompanied by eGFR of ≤45 ml/min/1,73 m². Empagliflozin is also associated with weight loss. (1)

In the ERO patients had a history of CV disease. (Appendix 1). It is not known how many of patients in clinical practice have a history of CV disease according to the ERO definition. In a publication by Norhammar et al patients with CVD was approximately 34 %. (2)However those data also included patients with atrial fibrillation and excluded patients with peripheral artery disease.

According to newly published Swedish guidelines by both the National board of Health and Welfare and the Medical Products Agency patients with type 2 diabetes and cardiovascular disease start treatment with Empagliflozin. (3) It is not known how many patients with T2DM and cardiovascular disease receive empagliflozin today.

## Research question and objectives

#### Research questions

- 1. Describe the prevalence of T2DM patients with established CVD according to ERO study definition in a Swedish population. (Appendix 1).
- 2. Describe the prevalence of established CVD according to ERO study definition in patients with T2DM who initiates treatment with empagliflozin.

### Objectives

### Primary objectives

- 1. To estimate the point prevalence of cardiovascular disease among persons with T2DM at 2017-12-31.
- 2. To estimate the prevalence of cardiovascular disease among persons with T2DM who initiates treatment with empagliflozin between 2015-01-01 and 2017-12-31

### Secondary objectives

- 1. Describe the T2DM patients with established CVD according to ERO study definition with respect to demographics and disease characteristics.
- 2. Describe the patients initiating with empagliflozin with respect to demographics and disease characteristics.

## Subject sets analyzed

Source population in the study

The broad study population will include patients with T2DM and at least one registration in the NDR (at any time from start of registry until 2017) and who are alive on 2015-01-01. Based on this population, the following two sub-populations will be identified, corresponding to each of the two research questions:

Table 1 Populations

| Population | Definition | Details | Data<br>source |
|---|---|---|---|
| Broad population | Patients with T2DM and at least one registration in the NDR (at any time from start of registry until 2017) and alive on 2015-01-01 | | NDR |
| Population 1 | Among the broader study population, those who are alive also on 2017-12-31 will be included. | | NDR |
| Population 2 | Among the broader study population, those | SPDR used to | NDR |

#### Index date

The index date for question 1 will be 2017-12-31. For question 2, the index date will be the date corresponding to the first collection of empagliflozin.

### Baseline and look back period

To characterize the study population, all information available during the look-back (pre-index) time period will be collected.

The look-back time period is defined as the time period ending on the day before the index date (Table 2).

Table 2 Data sources with look-back periods and total data collection periods

| Data source | Data holder | Look-back<br>period | Total data collection period |
|---|---|---|---|
| National diabetes register (NDR) | Centre of Registers,<br>Region Västra Götaland | 1 year | 1996-2017 |
| Swedish prescribed drug register (SPDR) | National Board of Health and Welfare | | 2015.01.01-<br>2017.12.31 |
| National patient register (NPR), both inpatient <sup>3</sup> and outpatient <sup>4</sup> registers | National Board of Health and Welfare | 1997-index<br>date (i.e. as<br>long as data<br>allows) | 1997-2017 |
| Cause of death register (CDR) | National board of health and welfare | Will be used<br>to establish the<br>broader<br>population and<br>population 2<br>(i.e to<br>establish that<br>patients are<br>alive) | 2017 |

| Variable | Definition | Details | Data<br>source |
|---|---|---|---|
| Established<br>CVD | Presence of at least one of the ICD10 codes as defined in appendix 1 | NPR introduced ICD10-codes in 1997, i.e. data from that year and later will be used | NPR<br>inpatient<br>and<br>outpatient |

## Initiation on Empagliflozin

 $Table\ 4\ Initiation\ of\ empagliflozin$ 

| Variable | Definition | Details | Data<br>source |
|---|---|---|---|
| Date for initiation of empagliflozin | The date for first collection of Empagliflozin (ATC code A10BK03) | Index date for<br>Question 2 | SPDR |

## Other variables

## Demographics and clinical baseline variables

Table 5 Demographics and other baseline variables

| Variable | Definition | Details | Data source |
|---|---|---|---|
| Age at index | Patient age at index. | Continuous | NDR |
| | Evaluated at the index date. | | |
| Sex | Patient sex. | Categorical: | NDR |
| | Evaluated at index date. | Female | |
| | | Male | |
| BMI | Patient BMI value at index date. | Continuous | NDR |
| | Evaluated at index date. | | |
| Smoking status | Patient smoking status at index date. | Categorical: | NDR |
| | Evaluated at the index date. | Yes | |

| | | No | |
|---|---|---|---|
| HbA1c value<br>(in mmol/mol) | Patient HbA1c measurement value at index date in mmol/mol. | Continuous | NDR |
| | Evaluated at the index date. | | |
| | Time difference between [index date] and [first type 2 diabetes diagnosis date]. | Continuous | NDR |
| date | Evaluated at the index date. | | |
| Systolic blood | Patient systolic blood pressure measurement | Continuous | NDR |
| pressure | value in mm Hg at then index date. | Continuous | NDK |
| | Evaluated at the index date. | | |
| Diastolic blood pressure | Patient diastolic blood pressure measurement value in mm Hg. | Continuous | NDR |
| | Evaluated at the index date. | | |
| Total cholesterol | Patient Total cholesterol measurement | Continuous | NDR |
| | Evaluated at the index date. | | |
| LDL | Patient LDL measurement value in mmol/L. | Continuous | NDR |
| | Evaluated at the index date. | | |
| HDL | Patient HDL measurement value in mmol/L. | Continuous | NDR |
| | Evaluated at the index date. | | |
| Triglyceride | Patient Triglyceride measurement value at index date in mmol/L. | Continuous | NDR |
| | Evaluated at the index date. | | |
| Creatinine | Patient Creatinine measurement | Continuos | NDR |
| | Evaluated at the index date. | | |
| Estimated glomerular filtration rate (eGFR) | Patient eGFR at index date estimate derived from serum creatinine measurement using the CKD-Epi equation: | Continuous | NDR |
| | eGFR (mL/min/1.73 $m^2$ ) = 141 x min(S <sub>cr</sub> /K,1) <sup>a</sup> x max(S <sub>cr</sub> /K,1) <sup>-1.209</sup> x 0.993 <sup>Age</sup> x 1.018 [if female]. | | |
| | a = -0.329 (females) or -0.411 (males). | | |
| | Evaluated at the index date. | | |
| Micro albuminurea | Evaluated at the index date. | Categorical: | NDR |

| | No | |
|---|---|---|
| Evaluated at the index date. | Categorical: | NDR |
| | Yes | |
| | No | |
| Evaluated at the index date. | | NDR |
| Evaluated at the index date. | | NDR |
| Evaluated at the index date. | | NDR |
| Evaluated at the index date. | | NDR |
| | Evaluated at the index date. Evaluated at the index date. Evaluated at the index date. | Evaluated at the index date. Categorical: Yes No Evaluated at the index date. Evaluated at the index date. Evaluated at the index date. |

## Planned analysis

### Summary of study populations identification

The identification process used to identify the study populations and subgroups will be summarized using population flowcharts including the following information:

- The total number of patients in the broad population (i.e. patients with T2DM and with at least one registration in the NDR and who are alive on 2015-01-01).
- The number of patients who are also alive on 2017-12-31 (the population for Question 1).
- The number of patients collecting Empagliflozin between 2015-01-01 and 2017-12-31 but who are not part of the broad population
- The number of patients in the broad population initiating Empagliflozin between 2015-01-01 and 2017-12-31 (the population for question 2)

### Main analysis

All analyses will be descriptive and no testing of hypotheses will be performed. The number and percentage of subjects with established CVD will be calculated and reported for both questions.

Variables in Table 5 will be descriptively reported for patients with established CVD within population 1 as well as for all patients in population 2.

Relating to question 2, the sub-group of patients initiating Empagliflozin during 2017 will be described with respect to prevalence of established CVD as well as the demographic and disease characteristics of Table 5.

## Data management

### Statistical software

The analysis and data management will be performed using SAS 9.4® or R 3.4.0.

R language is described in more details in report "R: Regulatory Compliance and Validation Issues: A Guidance Document for the Use of R in Regulated Clinical Trial Environments" (www.r-project.org/doc/R-FDA.pdf, read 21 December 2016).

### Quality control

Programs used in the data management and statistical analysis will be validated though independent review of the programming code, analysis data and output based on a risk assessment.

### References

- 1. Zinman et al. *Empagliflozin, cardiovascular outcomes, and mortality in Type 2 diabetes.* N Engl J Med 2015; 373:2117-2128
- 2. Norhammar et al. *Incidence, prevalence and mortality of type 2 diabetes requiring glucose-lowering treatment, and associated risks of cardiovascular complications: a nationwide study in Sweden, 2006–2013.* Diabetologia (2016) 59:1692–1701
- 3. Socialstyrelsen. 2017. *Nationella riktlinjer för diabetesvård*. Retrieved from http://www.socialstyrelsen.se/Lists/Artikelkatalog/Attachments/20633/2017-5-31.pdf